CLINICAL TRIAL: NCT02946346
Title: KINETICS AND ECOLOGY OF HUMAN PAPILLOMAVIRUS (HPV) GENITAL INFECTIONS IN YOUNG WOMEN
Brief Title: Kinetics and Ecology of Human Papillomavirus Genital Infections in Young Women
Acronym: PAPCLEAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to continue follow-up during the coronavirus epidemic
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL16_0149; 2016-A00712-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-08-22; First posted 2016-10-27 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2020-10

CONDITIONS: HPV Genital Infection (Primary Condition Studied); Bacterial Vaginosis; Chlamydiae Infection
Keywords: Human papillomaviruses; Clearance; Kinetics; Ecology; Bacterial vaginosis; Immune response; Microbiota
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal and blood sampling (Experimental)
  Interventions: Other: vaginal sampling

INTERVENTIONS:
Other: vaginal sampling

SUMMARY:
Most genital infections by human papillomaviruses (HPV) are asymptomatic or benign and clear within a few months or years. There infections are much less studies than chronic infections, even though they represent the main reservoir for the virus. The goal of this project is to decipher the kinetics of the virus and of the host immune response in acute HPV genital infections in your women. This will be performed by following women longitudinally and regularly in order to measure variations in virus load, immune cell count, cytokine concentration and antibody titers. The investigators will also investigate the interaction between these kinetics and host genetics and host vaginal microbiota

ELIGIBILITY:
Inclusion Criteria:

* Sexually active with at least one new partner over the last 12 months
* Subjects must be able and willing to give written informed consent
* Living in the 'agglomération de Montpellier'

Exclusion Criteria:

* History of cervical pathology
* Pregnant or intending to become pregnant soon (in the coming year)
* Infected by HIV
* Undergoing (or planning to undergo) heavy treatment (biotherapy, chemotherapy, immunosuppression)
* Participation in a clinical trial involving administration of drugswithin the last 4 weeks before the screening date

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Times series of HPV virus load in cervical smears measured by qPCR | from detection to clearance or persistence (i.e. 3 to 24 months)
  This time series will be used to calibrate a general model capturing HPV kinetics in genital acute infections in young women. At every time point, other measures such as temperature, vaginal pH, coinfections will be performed and women will fill-in detailed questionnaires about their every day life (vaccination status, antibiotic treatments, sexual activity) to control for co-factors. Virus genetics, host genetics (SNPs), immunophenotyping and microbiota will also be surveyed as cofactors.

SECONDARY OUTCOMES:
Times series of local innate and adaptive immune cell densities in cervical smears counted using Flow Cytometryor clearance) | from detection to clearance or persistence (i.e. 3 to 24 months)
  This time series will be used to calibrate a general model capturing HPV kinetics in genital acute infections in young women. At every time point, other measures such as temperature, vaginal pH, coinfections will be performed and women will fill-in detailed questionnaires about their every day life (vaccination status, antibiotic treatments, sexual activity) to control for co-factors. Virus genetics, host genetics (SNPs), immunophenotyping and microbiota will also be surveyed as cofactors.
Times series of vaginal cytokine densities measured using MesoScale Discovery technique | from detection to clearance or persistence (i.e. 3 to 24 months)
  This time series will be used to calibrate a general model capturing HPV kinetics in genital acute infections in young women. At every time point, other measures such as temperature, vaginal pH, coinfections will be performed and women will fill-in detailed questionnaires about their every day life (vaccination status, antibiotic treatments, sexual activity) to control for co-factors. Virus genetics, host genetics (SNPs), immunophenotyping and microbiota will also be surveyed as cofactors.
Times series of anti-HPV circulating antibody titers | from detection to clearance or persistence (i.e. 3 to 24 months)
  This time series will be used to calibrate a general model capturing HPV kinetics in genital acute infections in young women. At every time point, other measures such as temperature, vaginal pH, coinfections will be performed and women will fill-in detailed questionnaires about their every day life (vaccination status, antibiotic treatments, sexual activity) to control for co-factors. Virus genetics, host genetics (SNPs), immunophenotyping and microbiota will also be surveyed as cofactors.
Times series of the vaginal microbiota determined using 16S RNA and shotgun sequencing | from detection to clearance or persistence (i.e. 3 to 24 months)
  This time series will be used to calibrate a general model capturing HPV kinetics in genital acute infections in young women. At every time point, other measures such as temperature, vaginal pH, coinfections will be performed and women will fill-in detailed questionnaires about their every day life (vaccination status, antibiotic treatments, sexual activity) to control for co-factors. Virus genetics, host genetics (SNPs), immunophenotyping and microbiota will also be surveyed as cofactors.

CONTACTS AND LOCATIONS:
Locations (1):
- Pr Reynes, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tessandier N, Elie B, Boue V, Selinger C, Rahmoun M, Bernat C, Grasset S, Groc S, Bedin AS, Beneteau T, Bonneau M, Graf C, Jacobs N, Kamiya T, Kerioui M, Lajoie J, Melki I, Pretet JL, Reyne B, Schlecht-Louf G, Sofonea MT, Supplisson O, Wymant C, Foulongne V, Guedj J, Hirtz C, Picot MC, Reynes J, Tribout V, Tuaillon E, Waterboer T, Segondy M, Bravo IG, Boulle N, Murall CL, Alizon S. Viral and immune dynamics of genital human papillomavirus infections in young women with high temporal resolution. PLoS Biol. 2025 Jan 21;23(1):e3002949. doi: 10.1371/journal.pbio.3002949. eCollection 2025 Jan. PMID 39836629
- [Derived] Selinger C, Rahmoun M, Murall CL, Bernat C, Boue V, Bonneau M, Graf C, Grasset S, Groc S, Reynes J, Hirtz C, Jacobs N, Alizon S. Cytokine response following perturbation of the cervicovaginal milieu during HPV genital infection. Immunol Res. 2021 Jun;69(3):255-263. doi: 10.1007/s12026-021-09196-2. Epub 2021 Apr 30. PMID 33939124
- [Derived] Murall CL, Rahmoun M, Selinger C, Baldellou M, Bernat C, Bonneau M, Boue V, Buisson M, Christophe G, D'Auria G, Taroni F, Foulongne V, Froissart R, Graf C, Grasset S, Groc S, Hirtz C, Jaussent A, Lajoie J, Lorcy F, Picot E, Picot MC, Ravel J, Reynes J, Rousset T, Seddiki A, Teirlinck M, Tribout V, Tuaillon E, Waterboer T, Jacobs N, Bravo IG, Segondy M, Boulle N, Alizon S. Natural history, dynamics, and ecology of human papillomaviruses in genital infections of young women: protocol of the PAPCLEAR cohort study. BMJ Open. 2019 Jun 11;9(6):e025129. doi: 10.1136/bmjopen-2018-025129. PMID 31189673